CLINICAL TRIAL: NCT06097910
Title: Active Surveillance for Patients with Multifocal Ground-glass Nodules: a Prospective, Multi-center, Single-arm Trial (ECTOP-1021)
Brief Title: Surveillance for Multifocal GGNs
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director in the Department of Thoracic Surgery, FUSCC, Fudan University
Other Study IDs: ECTOP-1021
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-09

CONDITIONS: Lung Ground-glass Opacities; Active Surveillance
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observation
  Interventions: Procedure: Watchful waiting

INTERVENTIONS:
Procedure: Watchful waiting — Conduct thoracic computed tomography scans every 12 months. The decision regarding surgery is based on the surgeon's evaluation of radiologic follow-up. The reference resection criteria encompass: a) Any lesion that progresses to a tumor diameter larger than 2cm or has CTR greater than 0.25. b) Clinical Tumor, node, metastasis (TNM) stage upstaging.

SUMMARY:
This study is a single-arm, multi-center, phase III trial conducted under the Eastern Cooperative Thoracic Oncoloy Project (ECTOP) with the identification number ECTOP-1021. The primary objective of the study is to assess the overall survival of patients with multifocal ground-glass opacities by employing a active surveillance approach rather than opting for surgical resection.

DETAILED DESCRIPTION:
The trial aims to confirm the hypotheses that delaying surgery until GGO nodules exhibit progression or meet certain criteria offers a prognosis equivalent to those undergoing immediate surgical resection, potentially allowing many of these patients to avoid surgery altogether.

ELIGIBILITY:
Inclusion criteria Patients eligible for enrollment in the study are required to meet all the following criteria.

1. Demonstrates the following on thin-section computed tomography (TSCT) scan:

   1. Presence of three or more GGNs (bilateral lesions are permitted).
   2. All lesions have remained stable without regression or enlargement for at least 3 months.
   3. The dominant lesion (the lesion with the largest maximum tumor diameter) has a maximum tumor diameter >=0.6cm and <=2cm.
   4. CTR <=0.25 in all lesions.
   5. No lymph node with a diameter >1cm in the mediastinal view.
   6. Not adjacent to the pleura in dominant lesion and no sign of pleural retraction in any lesions.
2. Aged 18-75 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Has not previously undergo any anti-tumor drug or radiation therapy.
5. Written informed consent.

Exclusion criteria Patients will be excluded if they meet any of the following criteria.

1. History of any prior malignancies within the past 5 years.
2. History of lung surgery.
3. History of interstitial pneumonia, pulmonary fibrosis or other severe pulmonary diseases.
4. Presence of severe or uncontrolled diseases that may possibly reduce the 10-year life expectancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients who are willing to particiapte in the study and meet the inclusion and exculsion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2036-11-01 (Estimated); Study Completion 2036-11-01 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 5 years
  The event is defined as the death due to any causes.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The clinical data including patient characteristics and CT images.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within five years from the study end.
Access Criteria: Medical oncologists and surgeons who are interested in the study. Emails could be sent to the address below to obtain the shared data:
  hqchen1@yahoo.com

REFERENCES:
- [Derived] Wu H, Deng P, Fu F, Zhang Y, Chen H. Active surveillance for patients with multifocal ground-glass nodules: protocol of a prospective, multi-center, single-arm trial (ECTOP-1021). J Thorac Dis. 2025 Apr 30;17(4):2634-2639. doi: 10.21037/jtd-2024-1956. Epub 2025 Apr 28. PMID 40400915